CLINICAL TRIAL: NCT07084805
Title: Diabetes Inspired Culinary Education (DICE): An Innovative Approach to Type 1 Diabetes Management for At-Risk Youth With Type 1 Diabetes
Brief Title: Diabetes Inspired Culinary Education (DICE): Culinary Medicine Intervention for At-Risk Youth With Type 1 Diabetes
Acronym: DICE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: American Diabetes Association (Other); Rainbow Babies and Children's Hospital (Other); The Cleveland Clinic (Other); Breakthrough T1D (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20230091
Record Dates: First submitted 2025-07-23; First posted 2025-07-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
Keywords: Pediatrics; Culinary medicine; Teaching kitchen; Culinary nutrition
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Intervention Model Description: Waitlist Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receive DICE intervention during phase 1 while waitlist control arm receives usual clinical care.
  Interventions: Behavioral: Diabetes Inspired Culinary Education (DICE) - Phase 1
- Waitlist Control (Active Comparator): Receive DICE intervention during phase 2 while intervention arm receives usual clinical care.
  Interventions: Behavioral: Diabetes Inspired Culinary Education (DICE) - Phase 2

INTERVENTIONS:
Behavioral: Diabetes Inspired Culinary Education (DICE) - Phase 1 — The DICE intervention is a 10-lesson family-and community-based culinary nutrition and diabetes education program. Intervention Mapping, a protocol for developing theory- and evidence-based health promotion programs, was utilized to develop the DICE intervention. Rooted in the Social Cognitive Theory, the DICE intervention targets key personal, behavioral, and environmental constructs as mechanistic pathways for eliciting change in the consequential health outcomes of poor glycemic control in children and adolescents with type 1 diabetes.
  Arms: Intervention
Behavioral: Diabetes Inspired Culinary Education (DICE) - Phase 2 — The DICE intervention is a 10-lesson family-and community-based culinary nutrition and diabetes education program. Intervention Mapping, a protocol for developing theory- and evidence-based health promotion programs, was utilized to develop the DICE intervention. Rooted in the Social Cognitive Theory, the DICE intervention targets key personal, behavioral, and environmental constructs as mechanistic pathways for eliciting change in the consequential health outcomes of poor glycemic control in children and adolescents with type 1 diabetes.
  Arms: Waitlist Control

SUMMARY:
Diabetes Inspired Culinary Education (DICE) is an innovative family- and community-based culinary medicine intervention designed to mitigate racial/ethnic and socioeconomic status disparities in the treatment and health outcomes of at-risk youth with type 1 diabetes.

ELIGIBILITY:
Child Inclusion Criteria:

* Type 1 diabetes diagnosis for at least 12 months by study completion
* Poor glycemic control (1 HbA1c test results ≥ 7.0 % over the past 12 months or blood sugar levels > 155 mg/dL 3 or more times a week
* 8-14 years old
* English speaking

Caregiver Inclusion Criteria:

* Must be the primary caregiver of the participating child, (i.e., the individual who takes the lead role in helping the child manage their type 1 diabetes (e.g., monitoring blood sugars, planning meals/snacks, carbohydrate counting, etc.)
* 18 years of age or older
* English speaking

Child Exclusion Criteria:

* Not aged 8-14
* No demonstration of poor glycemic control
* Diagnosis of type 1 diabetes for less than 1 year by program completion
* Not English speaking

Caregiver Exclusion Criteria:

* Not the child's primary caregiver, (i.e., the individual who takes the lead role in helping the child manage their type 1 diabetes)
* Less than 18 years of age
* Not English speaking

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 9 months
  Blood glucose management

CONTACTS AND LOCATIONS:
Overall Officials: Catherine R McManus, PhD, RDN, LD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No